CLINICAL TRIAL: NCT07279389
Title: Comparative Study Between One-Shot Dilatation Versus Serial Dilatation Techniques for Access in Percutaneous Nephrolithotomy in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MS133/2022
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2022-08

CONDITIONS: Percutaneous Nephrolithotomy (PCNL); Renal Stone Disease
Keywords: Percutaneous Nephrolithotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients receiving renal dilatation by one-shot dilatation technique (Active Comparator): renal dilatation was done by one-shot dilatation technique using 30Fr Amplatz dilator directly over the central Alken rod.
  Interventions: Procedure: renal dilatation by one-shot dilatation technique
- Patients receiving renal dilatation by metallic telescopic dilators (Alken). (Active Comparator)
  Interventions: Procedure: renal dilatation by metallic telescopic dilators (Alken).
- Patients receiving renal dilatation by sequential fascial dilators (Amplatz). (Active Comparator)
  Interventions: Procedure: renal dilatation by sequential fascial dilators (Amplatz)

INTERVENTIONS:
Procedure: renal dilatation by one-shot dilatation technique — renal dilatation was done by one-shot dilatation technique using 30Fr Amplatz dilator directly over the central Alken rod.
  Arms: Patients receiving renal dilatation by one-shot dilatation technique
Procedure: renal dilatation by metallic telescopic dilators (Alken). — insertion of the Alken guide followed by a telescopic dilator between 9Fr to 30Fr, then an Amplatz sheath 30Fr was advanced over the dilator which was then removed, leaving the Amplatz sheath in the collecting system
  Arms: Patients receiving renal dilatation by metallic telescopic dilators (Alken).
Procedure: renal dilatation by sequential fascial dilators (Amplatz) — sequential renal dilatation with Amplatz dilator set was used
  Arms: Patients receiving renal dilatation by sequential fascial dilators (Amplatz).

SUMMARY:
This comparative study aims to compare and assess the safety, efficacy, outcome, feasibility, intraoperative and postoperative complications of one-shot dilatation versus serial dilatation techniques for access during percutaneous nephrolithotomy for management of renal stone disease in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years.
* Patients with renal stones which their size in maximum diameter is more than 2cm and indicated for percutaneous nephrolithotomy.
* Patients clinically fit for surgery.
* Patients with normal anatomy of urinary tract.
* Patients able to understand the procedure and accept to sign the informed consent.

Exclusion Criteria:

* Patients aged below 18 or above 70 years.
* Patients with renal stones which their size in maximum diameter is less than 2cm or contraindicated for endoscopic management.
* Patients with urinary tract infection, abnormal coagulopathy state or clinically unfit for surgery.
* Patients with nephrostomy tube in situ.
* Patients with more than single access tract.
* Patients undergoing simultaneous bilateral stone procedures.
* Patients with urinary tract abnormalities or history of renal transplantation.
* Renal insufficiency with serum creatinine above 3.0mg/dL
* Patients unable to understand the procedure or refuse to sign the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2022-08-27 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Mean Fluoroscopy time | From enrollment to the end of treatment at 8 weeks
Mean access time | From enrollment to the end of treatment at 8 weeks
Stone free rate | From enrollment to the end of treatment at 8 weeks
Hospitalization Period | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Arafa, Consultant, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Alken P, Hutschenreiter G, Gunther R, Marberger M. Percutaneous stone manipulation. J Urol. 1981 Apr;125(4):463-6. doi: 10.1016/s0022-5347(17)55073-9. PMID 7218439